CLINICAL TRIAL: NCT01356381
Title: A Single-center,Double-blind,Randomised,Placebo-controlled,Parallel-group Study to Assess the Effect of 24 Weeks of Treatment With Vildagliptin on Insulin Sensitivity and Its Underlying Mechanism in Patients With T2DM Treated With Metformin
Brief Title: Study to Assess the Effect of 24 Weeks of Treatment With Vildagliptin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLAF237A2389; 2006-004400-40 (EudraCT Number)
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes mellitus; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- vildagliptin (Experimental)
  Interventions: Drug: Vildagliptin
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin — Dosage 50mg b.i.d.
  Arms: vildagliptin
Drug: Placebo — 50mg bid
  Arms: Placebo

SUMMARY:
The study will demonstrate the effect of 24 weeks of treatment with vildagliptin compared to placebo on insulin sensitivity in patients with type 2 diabetes mellitus (T2DM) treated with metformin, assessed as glucose Rd (rate of glucose disposal) during a hyperinsulinemic euglycemic clamp.

ELIGIBILITY:
Inclusion Criteria:

1. Age in the range of 18-70 years.
2. Patients with T2DM, diagnosed at least 6 months prior to Visit 1, who have received metformin for at least 3 months and have been on a stable dose of at least 1000mg daily for a minimum of 4 weeks prior to Visit 1.
3. HbA1c ≤ 7.6% at Visit 1.
4. Body mass index (BMI) in the range of 22-38kg/m2 inclusive at Visit 1.

Exclusion Criteria:

1. Pregnant or nursing (lactating) women.
2. Patients with cardiac pacemakers or with metallic implants incompatible with magnetic resonance methodology.
3. Congestive heart failure requiring pharmacologic treatment. Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Measure: effect of treatment on insulin sensitivity, assessed as glucose Rd (rate of glucose disposal). | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Macauley M, Hollingsworth KG, Smith FE, Thelwall PE, Al-Mrabeh A, Schweizer A, Foley JE, Taylor R. Effect of vildagliptin on hepatic steatosis. J Clin Endocrinol Metab. 2015 Apr;100(4):1578-85. doi: 10.1210/jc.2014-3794. Epub 2015 Feb 9. PMID 25664602
- [Derived] Macauley M, Smith FE, Thelwall PE, Hollingsworth KG, Taylor R. Diurnal variation in skeletal muscle and liver glycogen in humans with normal health and Type 2 diabetes. Clin Sci (Lond). 2015 May 1;128(10):707-13. doi: 10.1042/CS20140681. PMID 25583442